CLINICAL TRIAL: NCT04749732
Title: Patient Education on a Quantified Supervised Home-based Exercise Therapy to Improve Walking Ability in Patients With Peripheral Arterial Disease and Intermittent Claudication: WalkingPad Protocol
Brief Title: Home-based Exercise Therapy for Patients With PAD
Acronym: WalkingPAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Hospitalar do Porto (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other); University of Trás-os-Montes and Alto Douro (Other); Institute for Systems and Computer Engineering, Technology and Science-INESC TEC (Unknown)
Responsible Party: Principal Investigator, Ivone Silva, Principal Investigator, Centro Hospitalar do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 069-DEFI/068-CES
Record Dates: First submitted 2021-02-03; First posted 2021-02-11 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Peripheral Arterial Disease (PAD); Intermittent Claudication
Keywords: Peripheral Arterial Disease; Arterial Occlusive Diseases; Vascular Diseases; Cardiovascular Diseases; Intermittent Claudication; Walking ability; Health-related Quality of Life; Home-based Exercise Therapy; Pervasive virtual assistant
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Arterial Occlusive Diseases; Vascular Diseases; Cardiovascular Diseases | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: This is a single-center three-arm parallel prospective, randomized controlled and superiority trial, with stratified random allocation, aiming to test the effectiveness of a Home-based Exercise Therapy (HbET) for claudicant patients to increase the Maximum Walking Distance (MWD), the Pain-free Walking Distance (PFWD) and the Functional Walking Distance (FWD). Patients will be assigned to one of three groups: an active control group (ACG); an experimental group 1 (GE1) and an experimental group 2 (EG2). All groups will have in common the prescription of a walking plan on a route defined by one of the team members through WalkingPAD web-platform and customized to the patient's home area. Participants from all three groups will undergo standard treatment for PAD and IC, according to the guidelines of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines.
Who Masked: Outcomes Assessor
Masking Description: Eligible participants will be randomly assigned to three groups in blocks of multiples of five and will be stratified according to i) age; and ii) mean walking distance at the baseline. This procedure will be performed using an online random number generator, by a researcher external to the team involved in the execution of this study, in order to ensure the concealment of the allocation of participants by the different groups. The participants will be blinded as to the group where they were allocated. After this procedure, it will not be possible to hide the group to which the patient belongs from the researcher who will carry out the psychological intervention and from the informatics engineer who will define the route of the walking plan. However, the outcome assessors (doctors, researchers, the clinical physiologist, and the exercise specialist) will be blinded to the allocation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WalkingPad plus Psychological Intervention - PsyWPad Group (Experimental): The participants in Experimental Group 1 will receive a prescription of an HBET consisting of a walking plan with a duration greater than 30 min per session, frequency of at least three sessions per week, use of near-maximal pain during training as claudication pain endpoint, with the support of a behavioral motivational intervention delivered by a health psychologist.
  Interventions: Behavioral: WalkingPad plus Psychological Intervention - PsyWPad Group
- WalkingPad plus Virtual Assistant - CyberWPad Group (Experimental): The participants in Experimental Group 2 will receive a prescription of an HbET consisting of a walking plan with a duration greater than 30 min per session, frequency of at least three sessions per week, use of near-maximal pain during training as claudication pain endpoint, with the support of a virtual assistant that will give motivational support.
  Interventions: Behavioral: WalkingPad plus Virtual Assistant - CyberWPad Group
- Paper WalkingPad group - PaperWPad Group (Active Comparator): The participants in the Active Control Group will receive a prescription of an HbET consisting of a walking plan with a duration greater than 30 min per session, frequency of at least three sessions per week, use of near-maximal pain during training as claudication pain endpoint, with the support of a behavioral motivational intervention delivered by a health psychologist.
  Interventions: Behavioral: WalkingPad group - Paper WPad Group

INTERVENTIONS:
Behavioral: WalkingPad plus Psychological Intervention - PsyWPad Group — The 24-week walking program will be monitored by the WalkingPAD application that will accompany the patient on their walks and record their adherence to the previously defined individual program. Motivational support for a behavioral intervention will include two face-to-face sessions and the following contacts will be made over the phone. The behavioral motivational intervention will follow the principles of 1) motivational interview, will be based on 2) Theory of self-determination, taking into account 3) components of the Transtheoretical Model of Change and the Theory of Planned Behavior.
  Other Names: Behavioral Change
  Arms: WalkingPad plus Psychological Intervention - PsyWPad Group
Behavioral: WalkingPad plus Virtual Assistant - CyberWPad Group — The 24-week walking program will be monitored by the WalkingPAD application, which will accompany the patient on their walks and record their adherence to the previously defined individual program. Motivational support will be provided by a virtual assistant through daily and on-the-spot interactions and through support and motivational messages.
  Other Names: Behavioral Change
  Arms: WalkingPad plus Virtual Assistant - CyberWPad Group
Behavioral: WalkingPad group - Paper WPad Group — The 24-week walking program will be supported by a printed prescription of an individualized HbET previously defined on the WalkingPAD platform. However, this group of patients will not have the support of an application to monitor and record adherence to the program. Motivational support for a behavioral intervention will include two face-to-face sessions and the following contacts will be made over the phone. The behavioral motivational intervention will follow the principles of 1) motivational interview, will be based on 2) Theory of self-determination, taking into account 3) components of the Trans-Theoretical Model of Change and the Theory of Planned Behavior.
  Other Names: Behavioral Change
  Arms: Paper WalkingPad group - PaperWPad Group

SUMMARY:
Cardiovascular disease represents a considerable economic burden to society and effective preventive measures are necessary. Patients with peripheral arterial disease (PAD) have a severe impairment of functional ability, namely in walking distance due to muscle ischemia defined as intermittent claudication (IC). The discomfort related to IC contributes to a sedentary lifestyle, decreasing physical fitness level, aggravating cardiovascular risk factors leading to disease deterioration. Exercise programs are an effective, low-cost, low-risk option compared with more invasive therapies for IC. Home-based exercise therapy (HBET) is structured, unsupervised, self-directed programs that take place in the personal setting of the patient rather than in a clinical setting. HBET program implementation is feasible and eliminates barriers such as transportation issues, proximity to clinics, and conflicts with occupational responsibilities. Even though these programs have shown to be effective at improving walking performance and distance, their results fall below those seen in Supervised Exercise Therapy (SET) programs. Thus, innovative home-based walking programs need to be developed in order to improve results and make exercise therapy available to a larger percentage of the population. The use of Information and communication technology (ICT) tools for self-monitoring is considered key to change long-term behavior. The WalkingPAD project aims to develop health technology assessment methods and evaluate personal health intervention strategies. Investigators intend to demonstrate the technical feasibility and economic viability of a personalized medicine application in real-life healthcare settings. This project intends to find evidence for three major questions: Does an M-health monitored home-based exercise program supported by a virtual assistant empowers commitment to exercise plan and allows remote control of plan accomplishment? Is it superior to an M-health monitored home-based exercise program supported by a behavioral motivational intervention, in increasing maximum walking distance? Is it superior to a self-monitoring exercise, with a specific self-designed walking plan in the residence area, in increasing maximum walking distance?

DETAILED DESCRIPTION:
Exercise training has been incorporated into current guidelines for the management of PAD. Multiple societal guidelines, including the American Heart Association Task Force on Clinical Practice Guidelines, Intersociety Consensus for the Management of PAD (TASC II), recommend supervised exercise therapy (SET) in the treatment of claudication symptoms in PAD. Consequently, the European Society of Cardiology proposes walking training as first-step therapy for claudicant patients before percutaneous or surgical options. Therefore, SET is the gold-standard for walking therapy in PAD patients. Although SET programs have proved to be more effective in increasing Maximum Walking Distance (MWD) and Pain-free Walking Distance (PFWD) compared with non-supervised exercise programs, they remain an underutilized tool and widespread implementation of SET is restricted by lack of facilities and funding. Home-based Exercise Therapy (HBET) has the advantage of providing a larger capacity of care, and in most cases, being feasibly close to the patients' home environment with reduced transport costs. Programs are self-directed with the guidance of healthcare providers that prescribe an exercise regimen similar to a supervised program. Thus, the primary goal of this study is to evaluate the effectiveness of an HBET program in increasing MWD, PFWD, and Functional Walking Distance (FWD). The study's primary outcomes will be MWD, PFWD, and FWD; secondary outcomes will be general and PAD-specific health-related quality of life (HRQoL) measures. A web platform and a mobile app will be created - WalkingPAD platform and app- allowing collaboration between several players, enhancing patient's compliance and accountability in their treatment strategy. Thus, an HBET will be prescribed to all the patients included in the study. The exercise prescription consists of: walking as the form of exercise, with a duration greater than 30 min per session, frequency of at least three sessions per week, using a near-maximal pain during training as claudication pain endpoint, and with a 6-month of duration. Participants will be randomized by three conditions - Active Control Group (ACG), an Experimental Group 1 (EG1), and an Experimental Group 2 (EG2) - stratified by age and MWD at baseline, and assessed at Time 1 (T1: before intervention), three months later (T2), and six months later (T3; follow-up). With WalkingPAD, investigators intend to demonstrate the technical feasibility and economic viability of a personalized medicine application in real-life healthcare settings and aspire to ensure coordination with national, regional, or local health authorities for dissemination and implementation of a new patient-centered, effective and low-cost therapeutic strategy.

Sample size calculation:

A total of 200 PAD patients with IC are expected to be recruited from the outpatient clinic of the Angiology & Vascular Surgery Department in CHUP-HSA in an attempt to account for the dropout rate and still achieve a large enough sample to obtain a 95% confidence interval. The minimum sample size of the total computerized sample for the 2 repeated measures (baseline and 3 months; and baseline and 6 months) was 54 participants, i.e. a minimum of 27 participants in each group (interventions groups and control group). The sample size was calculated for an effect size of 0.25, alfa of 0.05 and a power of 0,95 (1-beta) by the G*Power software.

Data Analysis:

Analyses of primary and secondary outcomes and process variables will be conducted on an intention-to-treat basis and all included participants will be analyzed as randomized.

Procedure:

Patients with PAD and IC, evaluated in the outpatient clinic of the Angiology & Vascular Surgery Department of CHUP-HSA between January and December of 2020 will be contacted by phone and invited to participate in the study. After obtaining oral consent by phone, a clinical, physical, hemodynamic and psychological evaluation will be scheduled at the hospital - Time 0 (T0 before assignment). In this assessment (T0), participants will sign a written consent and will be screened (1 hour +/-) to ascertain particular and specific exclusion and inclusion criteria.

Then, block randomization with four stratum will be performed. Stratum will be defined by age and mean walking distance at baseline. All patients will be informed of the goals, experimental procedures, risks, and benefits of the study. Signed informed consent from all patients will be obtained confirming adequate understanding of all information, voluntary decision and free from undue influence such as manipulation or coercion. The right of the recruited participants to change their minds and to abandon the investigation without penalty and with no obligation to justify shall be respected. All participants will have access to information about the new knowledge generated by the research to which they contributed. The privacy and confidentiality of patients' clinical data and respect for autonomy will be guaranteed. At Time 1 (T1), patients who meet the inclusion criteria (at T0) and accept to collaborate in this study will be (blind) allocated to one of the study's arms - ACG, EG1, or EG2, and evaluated with psychological and physical measures. Patients will be assessed after 3 months (T2) and six months (T3).

ELIGIBILITY:
Inclusion Criteria:

1. PAD with IC (Fontaine II ou Rutherford 1-3) due to atherosclerotic disease;
2. ABI below 0.9 at rest or below 0.73 after exercise (20% decrease);
3. Age range between 50 and 80;
4. MWD in treadmill test between 50 and 500 meters;

Exclusion Criteria:

1. Asymptomatic PAD;
2. Critical Ischemia (Fontaine III/IV or Rutherford 4-6);
3. Previous lower extremity vascular surgery, angioplasty, or lumbar sympathectomy;
4. Any condition other than PAD that limits walking;
5. Miocardial Infarction or Unstable Angina in the last 6 months;
6. Inability to obtain ABI measure because of non-compressible vessels;
7. Use of cilostazol and pentoxifylline initiated within 3 months before the investigation;
8. Active cancer, renal disease, or liver disease;
9. Severe chronic obstructive pulmonary disease (GOLD stage III/IV);
10. Severe congestive heart failure (NYHA class III/IV);

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Walking Distance (MWD) | Changes from before-assignment (T0 - treadmill and T1 - 6min walk test) to T2 (3 months), and to T3 (six-months)
  Maximum Walking Distance will be measured through the Treadmill Test and the 6 Minute Walk Test (6 MWT), in meters. The 6 MWT is a performance-based measure that evaluates the functional capacity of the individual to walk over a total of 6 min on a 100ft (≈30m) hallway, providing information regarding all the systems during physical activity.
Pain-free Walking Distance (PFWD) | Changes from before-assignment (T0 - treadmill and T1 - 6min walk test) to T2 (3 months), and to T3 (six-months)
  Pain-free Walking Distance (PFWD) will be measured through the Treadmill Test and the 6 Minute Walk Test (6 MWT), in meters. The 6 MWT is a performance-based measure that evaluates the functional capacity of the individual to walk over a total of 6 min on a 100ft (≈30m) hallway, providing information regarding all the systems during physical activity.
Functional Walking Distance (FWD) | Changes from before-assignment (T0 - treadmill and T1 - 6min walk test) to T2 (3 months), and to T3 (six-months)
  Functional Walking Distance (FWD) will be measured through the Treadmill Test and the 6 Minute Walk Test (6 MWT), in meters. The 6 MWT is a performance-based measure that evaluates the functional capacity of the individual to walk over a total of 6 min on a 100ft (≈30m) hallway, providing information regarding all the systems during physical activity.

SECONDARY OUTCOMES:
Physical Quality of Life | Changes from T0 (before-assignment) to T2 (3 months), and to T3 (six-months)
  Physical Quality of Life will be assessed through the Short-Form Health Survey (SF-36). Raw scores are transformed into a scale from 0 to 100. Higher results correspond to better physical quality of life. Higher results correspond to a better physical quality of life.
Mental Quality of Life | Changes from T0 (before-assignment) to T2 (3 months), and to T3 (six-months)
  Mental Quality of Life will be assessed through the Short-Form Health Survey (SF-36). Raw scores are transformed into a scale from 0 to 100. Higher results correspond to better mental quality of life. Higher results correspond to a better mental quality of life.
Vascular Disease specific Quality of Life | Changes from T0 (before-assignment) to T2 (3 months), and to T3 (six-months)
  Vascular disease-specific quality of Life will be assessed through the Vascular Disease-specific Quality of Life (VAsQoL-6). This is a specific measure for patients with PAD, assessing health-related quality of life in PAD. Scores range between 6 and 24, with higher results corresponding to a better quality of life associated with vascular disease.
Walking Impairment | Changes from T0 (before-assignment) to T2 (3 months), and to T3 (six-months)
  Walking impairment will be assessed through the Walking Impairment Questionnaire (WIQ) that assesses walking abilities in three domains:
  * distance (distances that the individual can walk) with scores ranging between 0 and 28, with higher results corresponding to greater distance;
  * speed (the speed that the individual can walk) with scores ranging between 0 and 16, with higher results corresponding to greater speed;
  * stairs (number of stairs that the individual can climb) with scores ranging between 0 and 12, with higher results corresponding to greater ability to climb stairs;

OTHER OUTCOMES:
Sociodemographic Data | T0 (before-assignment)
  The following socio-demographic data will be collected: gender; age; living environment; marital status; professional status; rural or urban areas of residence.
Clinical Data | T1 (before intervention) to T2 (3 months), and to T3 (six-months)
  The clinical data to collect will be: medical history, surgical history, chronic medication, lifestyle habits (alcohol and tobacco consumption, hours of sleep, and the number of meals per day).
Ankle-brachial-index (ABI) | T1 (before intervention) to T2 (3 months), and to T3 (six-months)
  The ABI measures the systolic pressures at the brachial artery, anterior tibial artery, and posterior tibial artery in the supine position in millimeters of mercury (mmHg), and will be assessed through a validated and certified Doppler device.
Transcutaneous Oxygen Pressure (TcPO2) | T1 (before intervention) to T2 (3 months), and to T3 (six-months)
  TcPO2 measures limb ischemia in millimeters of mercury (mmHg), and will be assessed through a validated and certified TcPO2 patient monitor.
Hand Strength | T1 (before intervention) to T2 (3 months), and to T3 (six-months)
  HGS measures and determines musculoskeletal function, weakness and disability in kilograms (kg), through a hand-held dynamometer.
Weight | T1 (before intervention) to T2 (3 months), and to T3 (six-months)
  Weight will be mesured in kilograms (kg), through a bioimpedance scale.
Height | [Time Frame: Changes from T1 (baseline) to T2 (3 months), and to T3 (six-months)]
  Height will be measured in Meters (mts), using a tape measure.
Body Mass Index | [Time Frame: Changes from T1 (baseline) to T2 (3 months), and to T3 (six-months)]
  Body mass index (kg/m2) will be measured through a bioimpedance scale.
Resting metabolism | [Time Frame: Changes from T1 (baseline) to T2 (3 months), and to T3 (six-months)]
  Resting metabolism of the patient will be measured in kilocalories (kcal) through a bioimpedance scale.
Body fat percentage | [Time Frame: Changes from T1 (baseline) to T2 (3 months), and to T3 (six-months)]
  Body fat percentage (%) will be measured through a bioimpedance scale.
Visceral fat level | [Time Frame: Changes from T1 (baseline) to T2 (3 months), and to T3 (six-months)]
  Visceral fat level (%) will be measured through a bioimpedance scale.
Skeletal muscle percentage | [Time Frame: Changes from T1 (baseline) to T2 (3 months), and to T3 (six-months)]
  Skeletal muscle percentage (%) will be measured through a bioimpedance scale.
Mental State | T0 (before-assignment)
  Mental state will be measured through the Mini-Mental State Examination (MMSE). This is a widely used test of cognitive function among the elderly, including tests of orientation, attention, memory, language, and visual-spatial skills. Higher results correspond to a better mental state.
Physical Performance | Changes from T0 (before-assignment) to T2 (3 months), and to T3 (six-months)
  Change in Physical performance will be measured through the International Physical Activity Questionnaire for the elderly (IPAQ_E) assesses self-reported moderate-to-vigorous physical activity (MVPA) and sedentary behavior (SB) in older adults, with scores ranging from 0 to indefinite minutes of physical activity per week and higher results correspond to a greater amount of physical activity performed. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity.
Anxiety Symptoms | Changes from T1 (baseline) to T2 (3 months), and to T3 (six-months)
  Anxiety symptoms will be measured through the Geriatric Anxiety Scale (GAS) assesses anxiety symptoms in older adults, with scores ranging from 0 to 5 and higher results correspond to more anxiety symptoms.
Depression Symptoms | [Time Frame: Changes from T1 (baseline) to T2 (3 months), and to T3 (six-months)]
  Depression symptoms will be measured through the Geriatric Depression Scale-5 (GDS) assesses depressive symptoms in older adults, with scores ranging from 0 to 5 and higher results correspond to more depression symptoms.
Stage of Change | Changes from T1 (baseline) to T2 (3 months), and to T3 (six-months)
  The Stage of Change will be measured through the Walking Motivation/Readiness for Change Questionnaire (WM/RCQ) which identifies the Stage of Change (SOC) in which participants are at the moment regarding walking training (Pre-contemplation, Contemplation, Preparation, Action, and Maintenance). Participants can only be in one stadium so the answer is exclusive to a single stadium (yes = 1; no = 0).
Locus of Causality | Changes from T1 (baseline) to T2 (3 months), and to T3 (six-months)
  Locus of causality will be measured through the Locus of Causality for Exercise Scale (LCES). This scale assesses the extent to which individuals feel that they freely choose to exercise rather than feeling that they have to for some reason. The response scale ranges from 3 to 18. Higher results indicate higher levels of autonomy (locus of causality internal).
Walking Planned Behavior | Changes from T1 (baseline) to T2 (3 months), and to T3 (six-months)
  Planned behavior will be assessed through the Walking Planned Behavior Questionnaire (WPBQ), which assesses intentions, attitudes, subjective norms, action and coping plans regarding walking. The response scale of ranges from 3 to 18. On the intentions scale, the score ranges between 2 and 10 points and higher scores indicate higher intention in do physical activity (walking); On the attitudes scale, the score ranges between 5 and 25 points and higher scores indicate a more positive the attitudes towards physical activity; On the subjective norms scale, the score ranges between 3 and 15 points, in which the higher the score, the higher is the perception of the importance attributed by other people to physical activity.
Illness representations | Changes from T1 (baseline) to T2 (3 months), and to T3 (six-months)
  Representations regarding PAD will be measured through the Illness Perception Questionnaire - Brief (IPQ-B). This assesses illness perceptions, with a response scale ranging from 0 to 10. Higher scores indicate more threatening perceptions regarding PAD.
Basic Psychological Need Satisfaction | Changes from T1 (baseline) to T2 (3 months), and to T3 (six-months)
  Basic Psychological Need Satisfaction will be assessed through the Psychological Need Satisfaction in Exercise Scale (PNSES). This scale assesses perceived psychological need satisfaction of the three basic psychological needs in the context of exercise (walking training): autonomy, competence, and positive relationship (relatedness). The response scale ranges from 12 to 60. Higher scores indicate more perceptions of psychological need fulfilment in exercise (walking).
Behavioral Regulation | Changes from T1 (baseline) to T2 (3 months), and to T3 (six-months)
  Regulation in Exercise will be measured through the Behavioral Regulation in Exercise Questionnaire (BREQ-3). This scale assesses the motivational regulations for walking training and the response scale ranges from 0 to 12 for each type of regulation. Higher results indicate higher levels of one of the following types of behavioral regulation: amotivation, external, introjected, identified, integrated, and intrinsic.
Cost-effectiveness of home-based exercise Vs. clinical-base exercise | At 6 months
  Compare cost-effectiveness analysis of HBET Control Vs. HBET with motivational support Vs. HBET with a virtual assistant. The outcome measure will be cost per quality adjusted life year (QALY)

CONTACTS AND LOCATIONS:
Overall Officials: Ivone Heitor, PhD, Principal Investigator — Centro Hospitalar do Porto
Locations (1):
- Centro Hospitalar do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, Collet JP, Czerny M, De Carlo M, Debus S, Espinola-Klein C, Kahan T, Kownator S, Mazzolai L, Naylor AR, Roffi M, Rother J, Sprynger M, Tendera M, Tepe G, Venermo M, Vlachopoulos C, Desormais I, Document Reviewers, Widimsky P, Kolh P, Agewall S, Bueno H, Coca A, De Borst GJ, Delgado V, Dick F, Erol C, Ferrini M, Kakkos S, Katus HA, Knuuti J, Lindholt J, Mattle H, Pieniazek P, Piepoli MF, Scheinert D, Sievert H, Simpson I, Sulzenko J, Tamargo J, Tokgozoglu L, Torbicki A, Tsakountakis N, Tunon J, Vega de Ceniga M, Windecker S, Zamorano JL. Editor's Choice - 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2018 Mar;55(3):305-368. doi: 10.1016/j.ejvs.2017.07.018. Epub 2017 Aug 26. No abstract available. PMID 28851596
- [Background] Al-Jundi W, Madbak K, Beard JD, Nawaz S, Tew GA. Systematic review of home-based exercise programmes for individuals with intermittent claudication. Eur J Vasc Endovasc Surg. 2013 Dec;46(6):690-706. doi: 10.1016/j.ejvs.2013.09.004. Epub 2013 Sep 11. PMID 24076079
- [Background] Aquino R, Johnnides C, Makaroun M, Whittle JC, Muluk VS, Kelley ME, Muluk SC. Natural history of claudication: long-term serial follow-up study of 1244 claudicants. J Vasc Surg. 2001 Dec;34(6):962-70. doi: 10.1067/mva.2001.119749. PMID 11743546
- [Background] Gerhard-Herman MD, Gornik HL, Barrett C, Barshes NR, Corriere MA, Drachman DE, Fleisher LA, Fowkes FG, Hamburg NM, Kinlay S, Lookstein R, Misra S, Mureebe L, Olin JW, Patel RA, Regensteiner JG, Schanzer A, Shishehbor MH, Stewart KJ, Treat-Jacobson D, Walsh ME. 2016 AHA/ACC Guideline on the Management of Patients With Lower Extremity Peripheral Artery Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2017 Mar 21;135(12):e686-e725. doi: 10.1161/CIR.0000000000000470. Epub 2016 Nov 13. PMID 27840332
- [Background] Berger JS, Ladapo JA. Underuse of Prevention and Lifestyle Counseling in Patients With Peripheral Artery Disease. J Am Coll Cardiol. 2017 May 9;69(18):2293-2300. doi: 10.1016/j.jacc.2017.02.064. PMID 28473134
- [Background] Collins TC, Lunos S, Carlson T, Henderson K, Lightbourne M, Nelson B, Hodges JS. Effects of a home-based walking intervention on mobility and quality of life in people with diabetes and peripheral arterial disease: a randomized controlled trial. Diabetes Care. 2011 Oct;34(10):2174-9. doi: 10.2337/dc10-2399. Epub 2011 Aug 26. PMID 21873560
- [Background] Duscha BD, Piner LW, Patel MP, Crawford LE, Jones WS, Patel MR, Kraus WE. Effects of a 12-Week mHealth Program on FunctionalCapacity and Physical Activity in Patients With PeripheralArtery Disease. Am J Cardiol. 2018 Sep 1;122(5):879-884. doi: 10.1016/j.amjcard.2018.05.018. Epub 2018 Jun 2. PMID 30049464
- [Background] Fakhry F, Spronk S, de Ridder M, den Hoed PT, Hunink MG. Long-term effects of structured home-based exercise program on functional capacity and quality of life in patients with intermittent claudication. Arch Phys Med Rehabil. 2011 Jul;92(7):1066-73. doi: 10.1016/j.apmr.2011.02.007. PMID 21704786
- [Background] Fokkenrood HJ, Bendermacher BL, Lauret GJ, Willigendael EM, Prins MH, Teijink JA. Supervised exercise therapy versus non-supervised exercise therapy for intermittent claudication. Cochrane Database Syst Rev. 2013 Aug 23;(8):CD005263. doi: 10.1002/14651858.CD005263.pub3. PMID 23970372
- [Background] Fokkenrood HJ, Lauret GJ, Scheltinga MR, Spreeuwenberg C, de Bie RA, Teijink JA. Multidisciplinary treatment for peripheral arterial occlusive disease and the role of eHealth and mHealth. J Multidiscip Healthc. 2012;5:257-63. doi: 10.2147/JMDH.S35779. Epub 2012 Oct 8. PMID 23093906
- [Background] Gardner AW, Parker DE, Montgomery PS, Blevins SM. Step-monitored home exercise improves ambulation, vascular function, and inflammation in symptomatic patients with peripheral artery disease: a randomized controlled trial. J Am Heart Assoc. 2014 Sep 18;3(5):e001107. doi: 10.1161/JAHA.114.001107. PMID 25237048
- [Background] Gardner AW, Parker DE, Montgomery PS, Scott KJ, Blevins SM. Efficacy of quantified home-based exercise and supervised exercise in patients with intermittent claudication: a randomized controlled trial. Circulation. 2011 Feb 8;123(5):491-8. doi: 10.1161/CIRCULATIONAHA.110.963066. Epub 2011 Jan 24. PMID 21262997
- [Background] Gardner AW, Poehlman ET. Exercise rehabilitation programs for the treatment of claudication pain. A meta-analysis. JAMA. 1995 Sep 27;274(12):975-80. PMID 7674529
- [Background] Golledge J, Singh TP, Alahakoon C, Pinchbeck J, Yip L, Moxon JV, Morris DR. Meta-analysis of clinical trials examining the benefit of structured home exercise in patients with peripheral artery disease. Br J Surg. 2019 Mar;106(4):319-331. doi: 10.1002/bjs.11101. Epub 2019 Feb 21. PMID 30791089
- [Background] Hageman D, Fokkenrood HJ, Gommans LN, van den Houten MM, Teijink JA. Supervised exercise therapy versus home-based exercise therapy versus walking advice for intermittent claudication. Cochrane Database Syst Rev. 2018 Apr 6;4(4):CD005263. doi: 10.1002/14651858.CD005263.pub4. PMID 29627967
- [Background] Harter M, Dirmaier J, Dwinger S, Kriston L, Herbarth L, Siegmund-Schultze E, Bermejo I, Matschinger H, Heider D, Konig HH. Effectiveness of Telephone-Based Health Coaching for Patients with Chronic Conditions: A Randomised Controlled Trial. PLoS One. 2016 Sep 15;11(9):e0161269. doi: 10.1371/journal.pone.0161269. eCollection 2016. PMID 27632360
- [Background] Harwood AE, Smith GE, Cayton T, Broadbent E, Chetter IC. A Systematic Review of the Uptake and Adherence Rates to Supervised Exercise Programs in Patients with Intermittent Claudication. Ann Vasc Surg. 2016 Jul;34:280-9. doi: 10.1016/j.avsg.2016.02.009. Epub 2016 Apr 25. PMID 27126713
- [Background] Khambati H, Boles K, Jetty P. Google Maps offers a new way to evaluate claudication. J Vasc Surg. 2017 May;65(5):1467-1472. doi: 10.1016/j.jvs.2016.11.047. Epub 2017 Mar 1. PMID 28259575
- [Background] Kivela K, Elo S, Kyngas H, Kaariainen M. The effects of health coaching on adult patients with chronic diseases: a systematic review. Patient Educ Couns. 2014 Nov;97(2):147-57. doi: 10.1016/j.pec.2014.07.026. Epub 2014 Aug 1. PMID 25127667
- [Background] Makris GC, Lattimer CR, Lavida A, Geroulakos G. Availability of supervised exercise programs and the role of structured home-based exercise in peripheral arterial disease. Eur J Vasc Endovasc Surg. 2012 Dec;44(6):569-75; discussion 576. doi: 10.1016/j.ejvs.2012.09.009. Epub 2012 Sep 30. PMID 23034408
- [Background] McDermott MM, Domanchuk K, Liu K, Guralnik JM, Tian L, Criqui MH, Ferrucci L, Kibbe M, Jones DL, Pearce WH, Zhao L, Spring B, Rejeski WJ. The Group Oriented Arterial Leg Study (GOALS) to improve walking performance in patients with peripheral arterial disease. Contemp Clin Trials. 2012 Nov;33(6):1311-20. doi: 10.1016/j.cct.2012.08.001. Epub 2012 Aug 7. PMID 23158112
- [Background] McDermott MM, Guralnik JM, Criqui MH, Ferrucci L, Zhao L, Liu K, Domanchuk K, Spring B, Tian L, Kibbe M, Liao Y, Lloyd Jones D, Rejeski WJ. Home-based walking exercise in peripheral artery disease: 12-month follow-up of the GOALS randomized trial. J Am Heart Assoc. 2014 May 21;3(3):e000711. doi: 10.1161/JAHA.113.000711. PMID 24850615
- [Background] McDermott MM, Guralnik JM, Criqui MH, Liu K, Kibbe MR, Ferrucci L. Six-minute walk is a better outcome measure than treadmill walking tests in therapeutic trials of patients with peripheral artery disease. Circulation. 2014 Jul 1;130(1):61-8. doi: 10.1161/CIRCULATIONAHA.114.007002. No abstract available. PMID 24982117
- [Background] McDermott MM, Polonsky TS. Home-Based Exercise: A Therapeutic Option for Peripheral Artery Disease. Circulation. 2016 Oct 18;134(16):1127-1129. doi: 10.1161/CIRCULATIONAHA.116.023691. No abstract available. PMID 27754945
- [Background] McDermott MM, Criqui MH, Greenland P, Guralnik JM, Liu K, Pearce WH, Taylor L, Chan C, Celic L, Woolley C, O'Brien MP, Schneider JR. Leg strength in peripheral arterial disease: associations with disease severity and lower-extremity performance. J Vasc Surg. 2004 Mar;39(3):523-30. doi: 10.1016/j.jvs.2003.08.038. PMID 14981443
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):e38-360. doi: 10.1161/CIR.0000000000000350. Epub 2015 Dec 16. No abstract available. PMID 26673558
- [Background] Muluk SC, Muluk VS, Kelley ME, Whittle JC, Tierney JA, Webster MW, Makaroun MS. Outcome events in patients with claudication: a 15-year study in 2777 patients. J Vasc Surg. 2001 Feb;33(2):251-7; discussion 257-8. doi: 10.1067/mva.2001.112210. PMID 11174775
- [Background] Nichols M, Townsend N, Scarborough P, Rayner M. Cardiovascular disease in Europe: epidemiological update. Eur Heart J. 2013 Oct;34(39):3028-34. doi: 10.1093/eurheartj/eht356. Epub 2013 Sep 7. PMID 24014390
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG, Rutherford RB; TASC II Working Group. Inter-society consensus for the management of peripheral arterial disease. Int Angiol. 2007 Jun;26(2):81-157. No abstract available. PMID 17489079
- [Background] Normahani P, Kwasnicki R, Bicknell C, Allen L, Jenkins MP, Gibbs R, Cheshire N, Darzi A, Riga C. Wearable Sensor Technology Efficacy in Peripheral Vascular Disease (wSTEP): A Randomized Controlled Trial. Ann Surg. 2018 Dec;268(6):1113-1118. doi: 10.1097/SLA.0000000000002300. PMID 28498233
- [Background] Parmenter BJ, Dieberg G, Smart NA. Exercise training for management of peripheral arterial disease: a systematic review and meta-analysis. Sports Med. 2015 Feb;45(2):231-44. doi: 10.1007/s40279-014-0261-z. PMID 25230780
- [Background] Rejeski WJ, Spring B, Domanchuk K, Tao H, Tian L, Zhao L, McDermott MM. A group-mediated, home-based physical activity intervention for patients with peripheral artery disease: effects on social and psychological function. J Transl Med. 2014 Jan 28;12:29. doi: 10.1186/1479-5876-12-29. PMID 24467875
- [Background] Rezvani F, Heider D, Harter M, Konig HH, Bienert F, Brinkmann J, Herbarth L, Kramer E, Steinisch P, Freudenstein F, Terhalle R, Grosse Y, Bock S, Posselt J, Beutel C, Reif F, Kirchhoff F, Neuschwander C, Loffler F, Brunner L, Dickmeis P, Heidenthal T, Schmitz L, Chase DP, Seelenmeyer C, Alscher MD, Tegtbur U, Dirmaier J. Telephone health coaching with exercise monitoring using wearable activity trackers (TeGeCoach) for improving walking impairment in peripheral artery disease: study protocol for a randomised controlled trial and economic evaluation. BMJ Open. 2020 Jun 4;10(6):e032146. doi: 10.1136/bmjopen-2019-032146. PMID 32503866
- [Background] Sakamoto S, Yokoyama N, Tamori Y, Akutsu K, Hashimoto H, Takeshita S. Patients with peripheral artery disease who complete 12-week supervised exercise training program show reduced cardiovascular mortality and morbidity. Circ J. 2009 Jan;73(1):167-73. doi: 10.1253/circj.cj-08-0141. Epub 2008 Nov 27. PMID 19039192
- [Background] Sampson UK, Fowkes FG, McDermott MM, Criqui MH, Aboyans V, Norman PE, Forouzanfar MH, Naghavi M, Song Y, Harrell FE Jr, Denenberg JO, Mensah GA, Ezzati M, Murray C. Global and regional burden of death and disability from peripheral artery disease: 21 world regions, 1990 to 2010. Glob Heart. 2014 Mar;9(1):145-158.e21. doi: 10.1016/j.gheart.2013.12.008. PMID 25432124
- [Background] Treat-Jacobson D, McDermott MM, Beckman JA, Burt MA, Creager MA, Ehrman JK, Gardner AW, Mays RJ, Regensteiner JG, Salisbury DL, Schorr EN, Walsh ME; American Heart Association Council on Peripheral Vascular Disease; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; and Council on Lifestyle and Cardiometabolic Health. Implementation of Supervised Exercise Therapy for Patients With Symptomatic Peripheral Artery Disease: A Science Advisory From the American Heart Association. Circulation. 2019 Sep 24;140(13):e700-e710. doi: 10.1161/CIR.0000000000000727. Epub 2019 Aug 26. PMID 31446770
- [Derived] Silva I, Moreira CS, Pedras S, Oliveira R, Veiga C, Moreira L, Santarem D, Guedes D, Paredes H. Effect of a monitored home-based exercise program combined with a behavior change intervention and a smartphone app on walking distances and quality of life in adults with peripheral arterial disease: the WalkingPad randomized clinical trial. Front Cardiovasc Med. 2023 Nov 22;10:1272897. doi: 10.3389/fcvm.2023.1272897. eCollection 2023. PMID 38075956
- [Derived] Silva I, Pedras S, Oliveira R, Veiga C, Paredes H. WalkingPad protocol: a randomized clinical trial of behavioral and motivational intervention added to smartphone-enabled supervised home-based exercise in patients with peripheral arterial disease and intermittent claudication. Trials. 2022 Apr 18;23(1):326. doi: 10.1186/s13063-022-06279-9. PMID 35436974